CLINICAL TRIAL: NCT07207161
Title: The Comparison of the Effects of a Single-Session Physiotherapy Intervention and Massage in Premature Infants: A Randomized Controlled Trial
Brief Title: Single-Session Physiotherapy Versus Massage in Premature Infants
Acronym: SPIM-Preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Seyma Atalar, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23090
Record Dates: First submitted 2025-09-11; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Preterm Infants
Keywords: Premature Infants; Physiotherapy; Infant Massage
MeSH Terms: conditions — Premature Birth | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model with three groups. Premature infants are randomly allocated to one of three arms: (1) Control group receiving routine neonatal care, (2) Massage group receiving infant massage, and (3) Physiotherapy group receiving a single-session physiotherapy intervention based on the Moyer-Mileur protocol.
Masking Description: This is an open-label study. Neither participants, care providers, investigators, nor outcome assessors are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Infants in this group will receive routine neonatal intensive care without any additional physiotherapy or massage intervention. This arm serves as the standard care control group.
- Massage Group (Experimental): Infants in this group will receive infant massage as an intervention. Massage will be performed by a trained physiotherapist following a standardized protocol. The purpose is to evaluate the effects of massage on physiological stability, weight gain, and overall development in premature infants.
  Interventions: Behavioral: Infant Massage
- Physiotherapy Group (Experimental): Infants in this group will receive a single-session physiotherapy intervention based on the Moyer-Mileur protocol. The intervention includes gentle range of motion and flexion-extension exercises designed to stimulate neuromuscular development in premature infants. The effects will be compared with those of massage and routine neonatal care.
  Interventions: Behavioral: Physiotherapy (Moyer-Mileur Protocol)

INTERVENTIONS:
Behavioral: Infant Massage — A standardized infant massage protocol applied by a physiotherapist, including gentle tactile stimulation to promote growth, relaxation, and neuromuscular development in premature infants.
  Arms: Massage Group
Behavioral: Physiotherapy (Moyer-Mileur Protocol) — A single-session physiotherapy intervention consisting of gentle range of motion and flexion-extension exercises following the Moyer-Mileur protocol to stimulate musculoskeletal and neuromotor development in premature infants.
  Arms: Physiotherapy Group

SUMMARY:
This study investigates the effects of a single-session physiotherapy intervention compared to massage in premature infants hospitalized in the neonatal intensive care unit. Premature babies are vulnerable to stress, pain, and sleep disturbances due to medical procedures and the intensive care environment. The study aims to evaluate whether physiotherapy or massage can reduce stress and pain, improve sleep, bilirubin levels, and cerebral oxygenation. Infants will be randomly assigned to three groups: control (routine care), massage, and physiotherapy (Moyer-Mileur protocol). The results will contribute to developing evidence-based interventions to support the health and development of premature infants

ELIGIBILITY:
Inclusion Criteria:

Preterm infants born between 20 and 37 gestational weeks

Apgar score ≥ 4 at the 5th minute after birth

Parental consent obtained for participation

Infants able to receive oxygen via CPAP (Continuous Positive Airway Pressure) or nasal prongs during the intervention if necessary

Exclusion Criteria:

Congenital anomalies or chromosomal abnormalities

Chronic medical conditions such as bronchopulmonary dysplasia

Intraventricular hemorrhage grade III or IV (IVH)

Necrotizing enterocolitis (NEC)

Asphyxia or seizures

Ages: 0 Days to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Neonatal Infant Stress Scale (NISS) | Pre-intervention to 30 minutes post-intervention
  Change in Neonatal Infant Stress Scale (NISS, range 0-2; higher scores indicate greater stress) before and after the intervention.
Change in Neonatal Infant Pain Scale(NIPS) | Pre-intervention to 30 minutes post-intervention
  Change in Neonatal Infant Pain Scale (NIPS, range 0-7; higher scores indicate more pain) before and after the intervention.
Change in Total Sleep Duration (Brief Infant Sleep Questionnaire) | Baseline (pre-intervention) and within 24 hours after the intervention
  Total sleep duration will be assessed using the Brief Infant Sleep Questionnaire (BISQ). Parents will be asked to report the infant's sleep pattern, and the total amount of time (in minutes) the infant sleeps during a 24-hour period will be recorded. The comparison will be made between pre-intervention and post-intervention data to evaluate whether the intervention has an effect on the infant's overall sleep time. A longer total sleep duration will be interpreted as an improvement in sleep quality.
Change in Number of Night Awakenings (Brief Infant Sleep Questionnaire) | Baseline (pre-intervention) and within 24 hours after the intervention
  Night awakenings will be assessed using the Brief Infant Sleep Questionnaire (BISQ). Parents will record the number of times the infant wakes up during the night within a typical 24-hour period. The data will be collected before and after the intervention to determine whether the procedure reduces the frequency of nighttime awakenings. A decrease in the number of awakenings will be considered as an indicator of improved sleep continuity and quality.
Change in Sleep Onset Latency (Brief Infant Sleep Questionnaire) | Baseline (pre-intervention) and within 24 hours after the intervention
  Sleep onset latency (the time it takes for the infant to fall asleep) will be measured using the Brief Infant Sleep Questionnaire (BISQ). Parents will report the average duration (in minutes) from when the infant is put to bed until the infant falls asleep. Comparisons will be made between pre-intervention and post-intervention values. A shorter sleep onset latency will be interpreted as a positive outcome, suggesting that the intervention may help infants fall asleep more quickly.

SECONDARY OUTCOMES:
Change in Oxygen Saturation (SpO₂-peripheral oxygen saturation) | 15 minutes before intervention, 5 minutes during intervention, and 15 minutes after intervention
  Oxygen saturation (SpO₂, measured in percentage) will be assessed to evaluate respiratory stability in premature infants during and after the intervention. Measurements will be recorded at three time points: (1) 15 minutes before the intervention (baseline), (2) at the 5th minute during the intervention, and (3) 15 minutes after the intervention. Higher oxygen saturation values (closer to 95-100%) will be considered favorable, indicating improved or maintained oxygenation.
Change in Heart Rate | 15 minutes before intervention, 5 minutes during intervention, and 15 minutes after intervention
  Heart rate (beats per minute) will be measured to assess physiological changes in premature infants following the intervention. Measurements will be taken at three distinct time points: (1) 15 minutes before the intervention (baseline), (2) during the intervention at the 5th minute, and (3) 15 minutes after the intervention. The purpose of this outcome is to determine whether the intervention has an effect on autonomic stability, as reflected by heart rate variability. A decrease in heart rate or stabilization within the normal neonatal range will be considered a favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Altuntaş Yılmaz, Study Director — Necmettin Erbakan University Nezahat Keleşoğlu Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Nezahat Keleşoğlu Faculty of Health Sciences, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.erbakan.edu.tr/tr/akademik-personel/5196-neslihan-altuntas-yilmaz